CLINICAL TRIAL: NCT07103005
Title: A 3-month Lifestyle Change Program's Impact on Body Composition, Resting Metabolic Rate, Food Intake and Health-related Quality of Life
Brief Title: Lifestyle Change: The Impact on Body Composition, Resting Metabolic Rate, Food Intake and Health-related Quality of Life
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VID Specialized University (Other)
Responsible Party: Principal Investigator, Hilde Trygstad, Section Leader, VID Specialized University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 761798; Reference number: 193383 (Other: VID Specialized University)
Record Dates: First submitted 2025-05-23; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Obesity and Overweight
Keywords: Body composition; healthy diet
MeSH Terms: conditions — Obesity; Overweight | interventions — Exercise; Diet

STUDY DESIGN:
Intervention Model Description: This study has a single group pre-post design. The intervention is an intensiv lifestyle intervention with physical activity focusing on muscle strength, and diet change focusing on more fruits, vegetables, proteins and fiber.
  Measurements were done before and after the intervention. Methods that were used were Bioelectrical impedance to measure body composition, questionires as RAND-36 to meassure HQoL, and DIGIKOST to measure diet.
  We also registered muscle- and fat mass with Dual-energy Ray Absorptiometry (DEXA) and whole-room indirect calorimet (WRIC).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A Commercial intensiv intervention with physical activity and diet. A single-group pre-post design (Experimental): All participants recieved the lifestyle intervention. Camparisons were made before and after the intervention.
  Body composition, Health realted quality of life and diet was registered before and after the intervention.
  Interventions: Procedure: Intensive behavioral change with physical activity and diet. A single-group pre-post design

INTERVENTIONS:
Procedure: Intensive behavioral change with physical activity and diet. A single-group pre-post design — The group of 43 participants recieved a lifestyle intervention, and was measurred before and after the intervention.
  The intervention was intensive physical activity with focus om muscle strength and dietary advice from dietition, with focus on more fruits, vegetables, proteins and fiber.
  Body composition was measurred using Bioelectrical impedance, DEXA and WRIC. Health related quality of life was measured using the questionnaire RAND-36, and diet was registered with the questionnaire DIGIKOST.
  Other Names: Diet; Physical activity; social support

SUMMARY:
In Norway, a significant proportion of the adult population is currently classified as overweight (~50%) or obese (~23%). Over the past four decades, there has been a significant rise in the prevalence of overweight and obesity in both children and adults. Obesity is associated with a higher risk of chronic diseases such as cardiovascular diseases, type 2 diabetes, respiratory disease, osteoarthritis and specific cancers. Consequently, leading to increased morbidity and reduction in life expectancy. A healthy lifestyle including meeting recommendations for diet and physical activity is considered beneficial the prevention of chronic diseases, and for quality of life. There is limited evidence on weight reduction programs implemented outside specialized healthcare services, however intensive lifestyle modifications have demonstrated promising effects on sustainable weight loss.

The Kickstart Program is a lifestyle program addressing weight reduction, changes in body composition and improved health-related quality of life (HRQoL) by integrating personalized dietary guidance and physical activity (PA) over a three, four or six-month period for registered participants, and can be considered an organized follow-up intervention. The participants receive close monitoring and support from clinical dietitians, physiotherapists and personal trainers. Unlike patients in specialized healthcare, Kickstart participants sign up and pay for it themselves, without any support from referrals or financial aid. This financial commitment is thought to make participants more motivated and facilitate compliance with the program. Recognizing the potential of programs like Kickstart to reduce healthcare costs by preventing lifestyle diseases, especially outside of specialized healthcare, shows why it is important to study how well they work.

The study's findings can be leveraged to assess the influence of lifestyle programs and enhance the support available to adults with obesity.

The study will tighten the knowledge gap concerning how an intervention of intensive dietary changes and PA specifically effects weight loss, FFM and HRQoL within a three-month timeframe.

The overall aim of the study is to investigate the effect of a combined diet and PA intervention for people with a BMI>25 kg/m² on body weight, body composition, RMR and HRQoL.

DETAILED DESCRIPTION:
In Norway, a significant proportion of the adult population is currently classified as overweight (~50%) or obese (~23%). Over the past four decades, there has been a significant rise in the prevalence of overweight and obesity in both children and adults. Obesity is associated with a higher risk of chronic diseases such as cardiovascular diseases, type 2 diabetes, respiratory disease, osteoarthritis and specific cancers. Consequently, leading to increased morbidity and reduction in life expectancy. A healthy lifestyle including meeting recommendations for diet and physical activity is considered beneficial the prevention of chronic diseases, and for quality of life. There is limited evidence on weight reduction programs implemented outside specialized healthcare services, however intensive lifestyle modifications have demonstrated promising effects on sustainable weight loss.

The Kickstart Program is a lifestyle program addressing weight reduction, changes in body composition and improved health-related quality of life (HRQoL) by integrating personalized dietary guidance and physical activity (PA) over a three, four or six-month period for registered participants, and can be considered an organized follow-up intervention. The participants receive close monitoring and support from clinical dietitians, physiotherapists and personal trainers. Unlike patients in specialized healthcare, Kickstart participants sign up and pay for it themselves, without any support from referrals or financial aid. This financial commitment is thought to make participants more motivated and facilitate compliance with the program. Recognizing the potential of programs like Kickstart to reduce healthcare costs by preventing lifestyle diseases, especially outside of specialized healthcare, shows why it is important to study how well they work.

Earlier studies have focused on the effect on body weight og body mass index (BMI). Because of the limitations with BMI, it is also important to study body composition. Body composition refers to the proportion of fat, muscle, bone, and other tissues that make up a person's body weight. It provides information about the distribution and relative proportions of body tissues, which can be important for evaluating overall health status, and progression of fitness during and after lifestyle change. Measurements of body composition can include body fat percentage (%), visceral fat, and fat free mass (FFM), including muscle mass that is the primary variable of interest in this study.

Resting metabolic rate (RMR) is the energy the body uses at rest to maintain vital functions. RMR is the main contributor to total energy expenditure, contributing up to 60-70 %. Other components of total energy expenditure is energy used from physical activity (20-30%) and lastly from the thermic effect of food (10%). Studies have demonstrated a decrease in RMR following weight loss, largely attributed to the loss of FFM, which plays a significant role in metabolic rate. It has been speculated that rapid weight loss induce metabolic adaptations resulting in greater than predicted decreases in RMR.

The concept of HRQoL is frequently utilized to assess how health status influences overall quality of life. Reported low HRQoL is typically found in individuals with multiple chronic conditions and low levels of PA.

In The Norwegian Healthy Life Centre Study by Samdal et al., the objective was to assess the impact of behavioral change interventions at Norwegian Healthy Life Centers on participants' physical activity six months after baseline. The study concluded that individuals with high socioeconomic status increased their physical activity more over the course of six months, but simultaneously consumed more unhealthy food. The intervention did not significantly influence dietary habits, but participants who attended the "good-food course" notably increased their consumption of healthy food. A follow-up study on HRQoL in 2020 revealed a positive association between physical activity and improved HRQoL. All HRQoL dimensions showed enhancement from baseline to the three-month follow-up, and these improvements were sustained at the 15-month follow-up.

By focusing on healthy lifestyle and weight reduction, valuable healthcare resources can be conserved, emphasizing the need for such programs outside specialized healthcare services. This also involves the individual's ability to cope and their overall quality of life. The study's findings can be leveraged to assess the influence of lifestyle programs and enhance the support available to adults with obesity.

The Kickstart program reveals a knowledge gap concerning how an intervention of intensive dietary changes and PA specifically effects weight loss, FFM and HRQoL within a three-month timeframe.

The overall aim of the study is to investigate the effect of a combined diet and PA intervention for people with a BMI>25 kg/m² on body weight, body composition, RMR and HRQoL.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 kg/m2

Exclusion Criteria:

* BMI< 25 kg/m2

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Bioelectircal impedance (BIA) | Base line to three months, and one year follow up
  Measurements of body composition i.e muscle mass was assessed by BIA
Dual-Energy X-Ray Absorptiometry (DEXA). | Base line to three months, and one year follow up
  Measurements of body composition i.e muscle mass was also assessed by DEXA
Resting energy expenditure (REE) | Base line to three months, and one year follow up
  REE was measured with indirect calorimetry
Questionnaire RAND 36-Item Short Form Health Survey (RAND-36) | Base line to three months, and one year follow up
  health related quality of life (HQoL) was assesed with RAND-36. RAND-36 has 36 questions with 8 dimentions. The scales are from 1-3 or 1-5. Low value estimates low scores.
Assessment of diet with Digikost questionnaire | Base line to three months, and one year follow up
  Diet change was measured with a validated digital food frequency questionnaire (FFQ):
  Digikost. The DIGIKOST-FFQ assesses data on single food items as well as food groups according to the Norwegian FBDG and the data is presented in grams per day. DIGIKOST-FFQ also presents variables of different food groups according to the recommendations (Norwegian food-based dietary guidelines)

CONTACTS AND LOCATIONS:
Locations (1):
- VID Specialized University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT07103005/Prot_000.pdf
  • Informed Consent Form (2024-04-17): https://cdn.clinicaltrials.gov/large-docs/05/NCT07103005/ICF_001.pdf